CLINICAL TRIAL: NCT05952791
Title: Laparoscopic Transabdominal Preperitoneal (TAPP) Groin Hernia Repair Using N-butyl-2-cyanoacrylate (LiquiBandFIX8®)for Mesh Fixation and Peritoneal Closure: Case Report About Extraperitoneal Hematoma
Brief Title: Case Report in Complications After Laparoscopic Transabdominal Preperitoneal Groin Hernia Repair Using LiquiBandFIX8®
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KeplerUH
Record Dates: First submitted 2023-06-07; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Groin Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surgery — Laparoscopic transabdominal preperitoneal (TAPP) groin hernia repair

SUMMARY:
This an a case report about management and proving the strenght and resistance of LiquiBandFIX8® using for peritoneal closure in a laparoscopic transabdominal preperitoneal groin hernia repair. The patient had anticoagulation due to a mechanical valvula and postoperatively the patient developed a huge hematoma extraperitoneally. Relaparoscopy war performed to identify the problem and check the peritoneal closure.

DETAILED DESCRIPTION:
This an a case report for proving the strenght and resistance of LiquiBandFIX8® using for peritoneal closure in a laparoscopic transabdominal preperitoneal groin hernia repair (TAPP). The patient had anticoagulation due to a mechanical valvula and postoperatively after TAPP the patient developed a huge hematoma extraperitoneally. The investigatorsperformed relaparoscopy for diagnostic and therapeutic reasons to check stop the bleeding and control the integrety of the peritoneal closure.

ELIGIBILITY:
Inclusion Criteria:

* Retrospective case report of one patient undergoing laparoscopic groin hernia repair

Exclusion criteria:

- not applicable (retrospective)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective case report of one patient
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Strongness of LiquiBandFIX8® | 2 weeks
  Mesh dislocation, mesh damage (yes/no)
Hemtoma | 2 weeks
  intraperitoneal blood (yes/no)
Strongness of LiquiBandFIX8® | 2 weeks
  peritoneal leakage, peritoneal damage (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Raab, MD, Principal Investigator — Kepler University Hospital Linz
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No